CLINICAL TRIAL: NCT02665000
Title: A Randomised Controlled Trial Evaluating the Effects of a Structured Training Program on the Learning Curve of Residents in the Field of Laparoscopic Surgery (STAR Trial)
Brief Title: Evaluating the Effects of a Structured Training Program on the Learning Curve of Residents in Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DSRB/2015/00944
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Laparoscopic Appendectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study arm: Structured training programme (Experimental): The participants in study arm will undergo 5 days training program in laparoscopic appendectomy using the Box and Wet Trainer as intervention. Each training session will take up to 2 hours. The participant will then be exposed to the standard training in current practice over 5 supervised cases of laparoscopic appendectomy.
  After the above training, they will be required to perform another 5 cases of laparoscopic appendectomy as performing surgeon under supervision by a trained surgeon. The operation will be recorded and graded based on a validated GOALS scoring system 6. The Primary Outcome will be the difference of the GOALS results between the 2 groups. Secondary outcomes will include OSAT score, patient outcome, residents' feedback score as well as conversion rates to open surgery.
  Interventions: Procedure: Structured training programme
- Control arm: non-training (No Intervention): Participant in study arm will not receive any additional training during the training week. The participant will then be exposed to the standard training in current practice over 5 supervised cases of laparoscopic appendectomy.
  They will be required to perform another 5 cases of laparoscopic appendectomy as performing surgeon under supervision by a trained surgeon. The operation will be recorded and then graded based on a validated GOALS scoring system 6

INTERVENTIONS:
Procedure: Structured training programme — Participants will undergo 5-days training sessions
  Other Names: Structured Training: Laparoscopic Appendectomy
  Arms: Study arm: Structured training programme

SUMMARY:
1.1 Aim The investigators wish to validate a structured training program for junior residents to enhance their learning curves in performing laparoscopic appendectomy.

1.2 Hypothesis To introduce a structured laparoscopic appendectomy training program and validate its efficacy with the validated GOALS scoring system.

DETAILED DESCRIPTION:
2. Background and clinical significance 2.1 Background The use of simulated training has been popularized for surgical techniques as it provides spatial and task oriented training which is vital for surgery. As more and more junior residents are performing laparoscopic appendectomy under supervision by registrars, the concern of patient safety of such early exposure without a prior structured training program is questioned. Furthermore, as these procedures are performed after office hours in our center, performance of this procedure by junior doctors may result in higher conversion rates according to a retrospective study done in our center.1 A recent leading article by Kordowicz et al stated the challenges and the importance of having validated simulator training for individual centers.2

2.2 Potential clinical significance The investigators propose that a validated training program will allow a safer training environment for junior residents. This will help to provide a standard laparoscopic training program that can be used for the training of future batches of surgical trainees coupled with improved learning curves and surgical techniques.

Studies done both locally and overseas have also shown that the presence of junior doctors in such operations can potentially increase operating time and poor surgical outcomes.3,4 Therefore, investigators also hope that with a validated training program for the residents, this can translate to improved patient outcomes and safety.

2.3 Potential benefits to the participants Direct benefit to the subjects include provision of a structured training program for participants randomized to Group A. Subjects in both groups will also receive critical assessment and feedback on their laparoscopic skills, thus contributing to the development of their surgical skills.

3. Methods Approach 3.1 Methodology A randomized controlled trial for junior surgical residents with less than 10 laparoscopic appendectomies' experience as first surgeon will be recruited. They will be randomized to either Group A or Group B (control).

3.2 Participants selection Junior surgical residents with less than 10 laparoscopic appendectomies' experience as first surgeon will be recruited. Up to 20 cases of laparoscopic appendectomies was shown to be the number required for a junior resident to become competent in the procedure.5

Residents who are in the post-graduate year 1(PGY-1) will be excluded from the study. This is as PGY-1 residents will be required to perform House Officer (HO) duties and as such do not participate in or perform any laparoscopic appendectomy procedures. Therefore, only surgical residents from PGY-2 to PGY-5 will be recruited.

3.3 Training Program Participants in Group A will undergo 5 days training program in laparoscopic appendectomy using the Box Trainer and Wet Trainer, whereas Group B will not receive any additional training during this week. Each training session will take up to 2 hours. Both groups will then be exposed to the standard training in current practice over 5 supervised cases of laparoscopic appendectomy.

After the above training, they will all be required to perform another 5 cases of laparoscopic appendectomy as performing surgeon under supervision by a trained surgeon. The operation will be recorded and then graded based on a validated GOALS scoring system 6 (Appendix A). The Primary Outcome will be the difference of the GOALS results between the 2 groups. Secondary outcomes will include OSAT score (Appendix B), patient outcome, residents' feedback score as well as conversion rates to open surgery.

3.4 Conducting the study The study subjects will be randomly assigned by a computer-generated randomization process to receive either the structured training program prior to standard current training practice (Group A) or only the standard current training practice (Group B, control).

A power calculation was performed to assess the number of participants required in the control and intervention groups. To detect a difference in GOALS score of 4, assuming an alpha of 0.05, a power of 0.80, the minimum number of subjects needed is 16.

All recruited residents will go through an aptitude test on the simulator to ensure comparability of the 2 groups prior to intervention.

Residents in Group A will receive up to 2 hours of supervised training by a trained surgeon per day for 5 days. The 2 hours will include a 30 minutes discussion on the training cases for the day, a 1 hour hands on practice with the Box Trainer as well as Wet Training followed by a 30 minutes feedback session.

Both groups will then be exposed to 5 cases of laparoscopic appendectomy with a trained surgeon as per current training practice.

The participants would then be graded for the next 5 cases of laparoscopic appendectomy that they perform. The assessment will include GOALS scoring by:

1. The supervising registrar
2. 2 consultant surgeons who will grade the resident's performance individually based on the video recording of the surgery

The study will be single-blinded as the assessors will not know which group each resident belong to. Blinding of residents would not be possible in this study. However, this would not affect the results of the primary outcome.

The laparoscopic appendectomies will be performed within a time period of 6 months as studies have shown that the effect of laparoscopic training do not persist beyond 6 months without any reinforcement.7

Feedback scores will be collated for all residents on completion of the study. The feedback scores will detail the level of confidence of the resident during the performance of the assessed cases and will be compared between the 2 groups.

A short summary of the process is as follows:

1. Consent of all subjects will be obtained
2. Pre-intervention aptitude assessment will be done for both Group A and B
3. 5 days of structured training program for subjects in Group A
4. Both groups will have a repeat aptitude test.
5. Both groups perform 5 training cases supervised by a trained surgeon, as of current training standards.
6. Assessment of subsequent 5 cases of laparoscopic appendectomies of subjects in both groups will be done by the senior surgeon assisting in each case as well as 2 independent consultant surgeons. This will be scored with the GOALS assessment.
7. Feedback scores on the level of confidence and competence in performing the 5 assessed cases will be collated for all subjects 3.5 Advantages of our study methodology Thus far, there have not been any locally validated training programs in literature. The studies on laparoscopic studies which have been conducted and validated overseas tend to focus on whether the use of a particular training tool (e.g. the use of laparoscopic stimulator, didactic lectures etc.) will be useful in improving the learning curves of the trainees.

Therefore, our research methodology is unique as it attempts to integrate the different training modalities that have been proven to improve the training curve into one seamless training program for the trainees. This seamless training will include didactic lectures as well as training on multiple different modalities, all of which has been shown in international journals to improve the learning curve of the trainees.

3.6 Potential limitations of the study Potential limitations will include

1. The difficulty level of each case of appendectomy will be different. This effect will be mitigated with randomization of the subjects to the 2 groups. In addition, the GOALS assessment takes into consideration the level of difficulty of the particular case and this will be reflected in the final score.
2. The amount of intervention from the registrar who is assisting in the surgery with the subject will differ. The GOALS assessment takes this into account and will allow the registrar to quantify the amount of assistance that was rendered intra-operatively. This will thus be reflected in the final score.

3.7 Potential harm/ hazard to participants and patients There are no potential risks to the patients in this study as the control arm residents will be receiving the same supervision as in our current day practice. All patients under this study will also go through the standard of care of laparoscopic appendectomy and no additional costs will be borne by the patients.

Similarly, for the participants in Group B (those who do not undergo the training program), the participants will not be in any form of disadvantage as they will still be undergoing the current training protocol.

3.8 Analyzing the data All the information that was recorded will be consolidated into a central form for each of the participants. The information obtained will be kept confidential and be kept in the office of the principal investigator (PI). Access to the information will only be given to the PI, co-PI and the collaborators.

The results of the trial will only be analyzed after completion of data collection. There will be no preliminary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Junior surgical residents with less than 10 laparoscopic appendectomies' experience as first surgeon will be recruited

Exclusion Criteria:

* Residents who are in the post-graduate year 1(PGY-1) will be excluded from the study

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The difference of the GOALS results between the 2 groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Choon Seng Chong, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] So JB, Chiong EC, Chiong E, Cheah WK, Lomanto D, Goh P, Kum CK. Laparoscopic appendectomy for perforated appendicitis. World J Surg. 2002 Dec;26(12):1485-8. doi: 10.1007/s00268-002-6457-7. Epub 2002 Sep 26. PMID 12297916
- [Background] Kordowicz AG, Gough MJ. The challenges of implementing a simulation-based surgical training curriculum. Br J Surg. 2014 Apr;101(5):441-3. doi: 10.1002/bjs.9370. Epub 2014 Feb 26. No abstract available. PMID 24615294
- [Background] Davis SS Jr, Husain FA, Lin E, Nandipati KC, Perez S, Sweeney JF. Resident participation in index laparoscopic general surgical cases: impact of the learning environment on surgical outcomes. J Am Coll Surg. 2013 Jan;216(1):96-104. doi: 10.1016/j.jamcollsurg.2012.08.014. Epub 2012 Sep 19. PMID 22999330
- [Background] Papandria D, Rhee D, Ortega G, Zhang Y, Gorgy A, Makary MA, Abdullah F. Assessing trainee impact on operative time for common general surgical procedures in ACS-NSQIP. J Surg Educ. 2012 Mar-Apr;69(2):149-55. doi: 10.1016/j.jsurg.2011.08.003. Epub 2011 Oct 2. PMID 22365858
- [Background] Gumbs AA, Hogle NJ, Fowler DL. Evaluation of resident laparoscopic performance using global operative assessment of laparoscopic skills. J Am Coll Surg. 2007 Feb;204(2):308-13. doi: 10.1016/j.jamcollsurg.2006.11.010. Epub 2006 Dec 27. PMID 17254935
- [Background] Schell SR, Flynn TC. Web-based minimally invasive surgery training: competency assessment in PGY 1-2 surgical residents. Curr Surg. 2004 Jan-Feb;61(1):120-4. doi: 10.1016/j.cursur.2003.08.011. PMID 14972187
- [Derived] Pang NQ, Chua HW, Kim G, Tan MY, Bin Abdul-Aziz MND, Xu RW, Chen E, Teo SC, Khoo NX, Lomanto D, Tai BC, So JB, Chong CS. Structured Training for Laparoscopic Appendectomy for Residents (STAR Trial)-A Randomized Pilot Study. J Surg Res. 2021 Dec;268:363-370. doi: 10.1016/j.jss.2021.06.073. Epub 2021 Aug 14. PMID 34399358